CLINICAL TRIAL: NCT03303729
Title: Influence of Carbohydrate on Amino Acid Absorption From Dietary Protein
Brief Title: Influence of Carbohydrate on Amino Acid Absorption From Dietary Protein (ICADP)
Acronym: ICADP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: University of Birmingham (Other)
Responsible Party: Principal Investigator, Lars Holm, PhD, MSc, Bispebjerg Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-17017363
Record Dates: First submitted 2017-10-03; First posted 2017-10-06 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Muscle Protein Synthesis; Amino Acid
Keywords: Carbohydrate; Cluster Dextrin; Exercise training; Protein supplement
MeSH Terms: interventions — Long-Term Synaptic Depression; Glucose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meat hydrolysate & Cluster Dextrin (Experimental): Meat hydrolysate containing 25g of protein given together with 75 grams of Cluster Dextrin.
  Interventions: Dietary Supplement: Meat Hydrolysate; Dietary Supplement: Cluster Dextrin
- Meat hydrolysate & placebo (Active Comparator): Meat hydrolysate containing 25g of protein given together with 75 grams of Glucose.
  Interventions: Dietary Supplement: Meat Hydrolysate; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Meat Hydrolysate — 25 grams of meat hydrolysate to maximally stimulate protein synthesis.
Dietary Supplement: Cluster Dextrin — 75 grams of Cluster Dextrin
  Other Names: CAS no.: 9050-36-6; Glico Nutrition Co., Ltd.
  Arms: Meat hydrolysate & Cluster Dextrin
Dietary Supplement: Placebo — 75 grams of Glucose
  Other Names: Glucose
  Arms: Meat hydrolysate & placebo

SUMMARY:
10 young males will be recruited to participate in a randomized double blinded crossover study to investigate the influence of concomitant intake of two different types of carbohydrate with protein hydrolysate on the absorption kinetics of protein-derived amino acids and the impact on myofibrillar protein synthesis. During the trial days the subjects will perform a bout of whole body resistance exercise and ingest a supplement of meat hydrolysate labeled with D5-phenylalanine together with randomized and double blinded type of carbohydrate consisting of either glucose or cluster dextrin.

The primary outcome is the time to obtain peak concentration of D5-phenylalanine after intake of meat hydrolysate with either glucose or cluster dextrin.

Hypotheses:

I) The cluster dextrin will increase the absorption of the amino acids from the meat hydrolysate, and thereby result in a faster rise and a higher peak in plasma amino acid concentration in the postprandial period.

II) The meat hydrolysate will increase the protein synthesis rate to a higher extent when combined with cluster dextrin than with glucose.

ELIGIBILITY:
Inclusion Criteria:

* young healthy adults,
* organised sport/training 1-3 times per week

Exclusion Criteria:

* Subject younger than 18 years or above 30 years
* BMI > 30
* Chronic medical diseases: active cancer, renal diseases, metabolic diseases like diabetes mellitus.
* Physical inactivity. Subjects must participate in systematized weekly exercise 1-3 times per week.
* Participating in systematized exercise more than 3 times per week.
* Vegetarian.
* Participating in a special diet which deviates from the standard of young adults.

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2017-11-24 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2018-02-23 (Actual)

PRIMARY OUTCOMES:
Protein hydrolysate amino acid label time to peak appearance in plasma | From hour 0 to hour 3
  Difference between the time to peak of protein-derived D5-phenylalanine amino acid appearance in the plasma

SECONDARY OUTCOMES:
Myofibrillar protein fractional synthesis rate response to protein and carbohydrate intake after a whole body resistance exercise | from hour 0,5 to hour hour 1. From hour 1 to hour 3. From hour 0,5 to hour 3.
  Difference between myofibrillar protein fractional synthesis rate after meat hydrolysate with either 75 grams of Cluster Dextrin or Clucose.
Protein hydrolysate amino acid label area under the concentration curve in plasma | From hour 0 to hour 3
  Difference between the area under the concentration curve of protein-derived D5-phenylalanine amino acid appearance in the plasma
Insulin concentration | From hour 0 to hour 3
  Difference between insulin concentrations after intake of the two carbohydrate types.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob L. Bülow, MD, Principal Investigator — Bispebjerg Hospital; Lars Holm, Prof., Principal Investigator — University of Birmingham; Michael Kjaer, MD, prof., Principal Investigator — Bispebjerg Hospital; Sofus Sølyst, stud.med., Principal Investigator — University of Copenhagen; Mikkel Jensen, Stud.scient., Principal Investigator — University of Copenhagen
Locations (1):
- Bispebjerg Hospital, Copenhagen, Copenhagen NV, Denmark

REFERENCES:
- [Derived] Nishimura Y, Jensen M, Bulow J, Thomsen TT, Arimitsu T, van Hall G, Fujita S, Holm L. Co-ingestion of cluster dextrin carbohydrate does not increase exogenous protein-derived amino acid release or myofibrillar protein synthesis following a whole-body resistance exercise in moderately trained younger males: a double-blinded randomized controlled crossover trial. Eur J Nutr. 2022 Aug;61(5):2475-2491. doi: 10.1007/s00394-021-02782-y. Epub 2022 Feb 19. PMID 35182194